CLINICAL TRIAL: NCT06311812
Title: Retrospective Review on Uterovaginal Anomalies
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, YEUNG Yat Ka ESTHER, Clinical Tutor (honorary), Chinese University of Hong Kong
Other Study IDs: CREC 2023.683
Record Dates: First submitted 2024-01-18; First posted 2024-03-15 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Abnormalities Uterine; Vaginal Abnormality
MeSH Terms: conditions — Uterine Anomalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Review of surgical outcomes of patient who have undergone surgery for uterovaginal anomalies. Case notes of patients would be reviewed and data would be gathered for statistical analysis.

DETAILED DESCRIPTION:
Uterovaginal anomalies are congenital malformations of the female reproductive tract, including hymenal, vaginal, cervical and uterine anomalies. The incidence could be as high as 7% in females1. These anomalies can occur alone or in association with other anomalies such as renal anomalies.

There could be variable consequences from these malformations, some are asymptomatic while some may have various symptoms.

It is important to be aware that obstructive uterovaginal anomalies, examples including imperforated hymen and obstructive hemivagina and ipsilateral renal anomaly (also known as OHVIRA), may present after puberty, with symptoms including amenorrhoea, dysmenorrhea, pelvic pain etc. These are conditions that should be managed. Patient may require interventions. Surgery is the principal management for obstructive anomalies, dependent on the types of obstruction. Types of surgeries ranges from simple surgical procedures to complex surgeries that require multidisciplinary input.

Post-operatively patients should be offered follow up for monitoring in view of the risk of stenosis that may require ongoing dilation or additional surgical management.

There are limited studies on the post-operative outcomes for uterovaginal anomalies, so this study aims at reviewing and comparing the different outcomes after initial surgery.

This is a retrospective observational study. Electronic and paper clinical records of all patients who attended the Prince of Wales Hospital, Alice Ho Miu Ling Nethersole Hospital and North District Hospital with the diagnosis of uterovaginal anomaly will be reviewed, data collected will be input and analyzed using different statistical analysis tools. Data between 1.1.2000 and 31.12.2023 will be reviewed retrospectively. No human subject will be recruited.

The aim of the study is to reviewing and comparing the different outcomes after surgery for patients who had uterovaginal anomalies

ELIGIBILITY:
Inclusion Criteria:

* All patients who attended the Prince of Wales Hospital with the diagnosis of uterovaginal anomaly since 2000

Exclusion Criteria:

* Nil

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All patients who attended the Prince of Wales Hospital, Alice Ho Miu Ling Nethersole Hospital and North District Hospital with the diagnosis of uterovaginal anomaly between 1.1.2000 and 31.12.2023.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of re-stenosis | 1 year after operation
  Patient record will be reviewed. Number of patients need re-stenosis after surgical treatment for obstructive uterovaginal anomalies will be counted.
Incidence of re-operation | 1 year after operation
  Patient record will be reviewed. Number of patients need re-operation after surgical treatment for obstructive uterovaginal anomalies will be counted.
Number of patients with normal menstruation after operation | 1 year after operation
  Menstruation status will be reviewed in post-operation follow up. Number of patients with normal menstruation after surgical treatment for obstructive uterovaginal anomalies will be counted.
Number of patients with sexual intercourse after operation | 1 year after operation
  Sexual status will be asked in post-operation follow up. Number of patients with sexual intercourse after surgical treatment for obstructive uterovaginal anomalies will be counted.
Number of patients with post-operative infection | 1 year after operation
  Patient record will be reviewed. Number of patients with post-operative infection will be counted.
Number of patients with pregnancy after operation | 1 year after operation
  Pregnancy status will be reviewed. Number of patients with ultrasound confirmed pregnancy after operation will be counted.

SECONDARY OUTCOMES:
Background demographics affecting post-operative outcomes for patients with uterovaginal anomalies | 1 year after operation
  Background demographics including age at diagnosis, age at operation, difference in age between menarche and diagnosis/ operation, history of previous abdominal or reproductive tract surgery, menstrual cycle will be reviewed.
  Categorical data will be analyzed with Chi square or Fisher's exact test. Continuous data will be analyzed with t test and ANOVA test. The significance level is set at 0.05.
Number of participants with Pre-operative factors affecting post-operative outcomes | 1 year after operation
  Pre-operative factors including presentation at diagnosis, laterality of hematocolpos, thickness and size of septum, distance of septum to perineum, obstructed longitudinal septum axis and the type of renal anomaly will be reviewed.
  Categorical data will be analyzed with Chi square or Fisher's exact test. Continuous data will be analyzed with t test and ANOVA test. The significance level is set at 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong